CLINICAL TRIAL: NCT02474927
Title: Combination Therapy With the Proteasome Inhibitor Carfilzomib for the Antibody-Mediated Rejection Diagnosis in Lung Transplantation Trial (PICARD-Lung)
Brief Title: Combination Therapy With Carfilzomib for the Antibody-Mediated Rejection Diagnosis in Lung Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John F. McDyer, MD (Other)
Responsible Party: Sponsor-Investigator, John F. McDyer, MD, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO15010152
Record Dates: First submitted 2015-05-21; First posted 2015-06-18 (Estimated); Results first posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Lung Transplant Rejection
Keywords: antibody-mediated rejection; lung transplant; Carfilzomib
MeSH Terms: interventions — carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carfilzomib Treatment Arm (Experimental): Carfilzomib will be administered at a dose of 20 mg/m2 on two consecutive days, each week for three weeks (Days 1 2, 8, 9, 15, and 16) to constitute one therapeutic cycle. Carfilzomib may be administered for 1-2 complete cycles in the study.
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib will be used in combination with the conventional therapy (plasma exchange and intravenous immunoglobulins)
  Other Names: Kyprolis

SUMMARY:
The clinical trial is a Phase II open label, single-arm pilot study to evaluate the safety and efficacy of combination therapy with carfilzomib, plasma exchange and intravenous immunoglobulins for AMR after lung transplantation and elucidate important clinical and immunologic phenotypes and mechanisms associated with these outcomes.

DETAILED DESCRIPTION:
The main objective of the proposed clinical investigation is to evaluate the effects of carfilzomib in addition to conventional therapy on short-term outcomes after the diagnosis of antibody-mediated rejection in lung transplant recipients. In this study, Carfilzomib will be administered at a dose of 20 mg/m2 on two consecutive days, each week for three weeks (Days 1 2, 8, 9, 15, and 16) to constitute one therapeutic cycle. Carfilzomib may be administered for 1-2 complete cycles in the study. Patients will be followed for the duration of their hospital admission after enrollment. Post treatment follow-up will also occur on Days 42 and 90.

ELIGIBILITY:
Inclusion Criteria:

* Adult lung transplant recipients ≥ 18 years of age who meet the diagnostic criteria for AMR and who have underwent PFT testing unless intubated and transbronchial biopsy prior to enrollment.

Exclusion Criteria:

* Direct contraindications or previous intolerances to any component of the standard of care regimen including PLEX, 5% human albumin, 5% gammagard S/D or 10% gammagard liquid
* Leukopenia
* Neutropenia
* Thrombocytopenia
* Known Child-Pugh B/C cirrhosis
* Total bilirubin > 4
* ALT > 90
* Known systolic heart failure with LVEF < 40%
* Known pulmonary hypertension
* Any uncontrolled comorbid condition
* Pregnant women
* Breastfeeding women
* Ongoing bacterial or fungal or viral infection that is life-threatening
* Active cytomegalovirus disease
* Active varicella zoster infection
* Previous intolerance to carfilzomib
* Concurrent use of another proteasome inhibitor (e.g., bortezomib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2021-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McDyer, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carfilzomib Treatment Arm
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 48 [21 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Decrease in Titer of One or More DSA (Either Reduced MFI or Absence of DSA on Same Dilution)
Description: Number of Participants with a Decrease in titer of one or more DSA (either reduced MFI or absence of DSA on same dilution).
Time Frame: Day 1 to Day 42
Population: Decrease in titer of one or more DSA (either reduced MFI or absence of DSA on same dilution)
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 22
Participants | 17

2. Primary Outcome: Number of Participants With a Decrease in DSA Titer
Description: Number of Participants with a Decrease in DSA Titer.
Time Frame: Day 1 to Day 42
Population: Change in DSA Titer (Titer Decreased) [6 not evaluable]
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 16
Participants | 13

3. Primary Outcome: Number of Participants With an Absence of One or More Previously Positive DSA on Cq1 Assay
Description: Number of Participants with an Absence of one or more previously positive DSA on Cq1 assay.
Time Frame: Day 1 to Day 42
Population: Absence of one or more previously positive DSA on Cq1 assay [14 not evaluable]
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 8
Participants | 5

4. Secondary Outcome: Number of Participants With a Decrease in Titer of One or More DSA (Either Reduced MFI or Absence of DSA on Same Dilution)
Description: as for outcome 1
Time Frame: Day 1 to Day 90
Population: Decrease in titer of one or more DSA (either reduced MFI or absence of DSA on same dilution)[2 not evaluable]
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 20
Participants | 17

5. Secondary Outcome: Number of Participants With a Decrease in DSA Titer
Description: Number of Participants with a Decrease in DSA Titer.
Time Frame: Day 1 to Day 90
Population: Change in DSA Titer (Titer Decreased) [9 not evaluable]
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 13
Participants | 10

6. Secondary Outcome: Number of Participants With an Absence of One or More Previously Positive DSA on Cq1 Assay
Description: Number of Participants with an Absence of one or more previously positive DSA on Cq1 assay.
Time Frame: Day 1 to Day 90
Population: Absence of one or more previously positive DSA on Cq1 assay [12 not evaluable]
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 10
Participants | 6

7. Secondary Outcome: Absolute Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: Absolute change in forced expiratory volume in 1 second (FEV1)
Time Frame: Day 1 to Day 42
Measure: Median (Full Range); unit: FEV1%
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 22
FEV1%
  Baseline | 1.77 [0.80 to 2.83]
  Day 42 | 1.93 [1.06 to 3.22]
Statistical Analysis 1: Comparison: Carfilzomib Treatment Arm; Test type: Other — Descriptive (Pre-Post); p = 0.36, Wilcoxon Signed Rank

8. Secondary Outcome: Absolute Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: Absolute Change in Forced Expiratory Volume in 1 Second (FEV1)
Time Frame: Day 1 to Day 90
Measure: Median (Full Range); unit: Median FEV1 value
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 22
Median FEV1 value
  Baseline | 1.77 [0.80 to 2.83]
  Day 90 | 2.09 [0.71 to 3.65]
Statistical Analysis 1: Comparison: Carfilzomib Treatment Arm; Test type: Other — Descriptive (pre-post); p = 0.16, Wilcoxon Signed Rank

9. Secondary Outcome: Presence or Absence of Pathologic Changes Consistent With AMR on Transbronchial Biopsy
Description: Presence or absence of pathologic changes consistent with AMR on transbronchial biopsy
Time Frame: Day 1 to Day 42
Population: Unable to calculate at dates specified at this time. Re-biopsy of patients is not routinely completed. Research biopsy was not part of the protocol.
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 0

10. Secondary Outcome: Patient Death Attributable to AMR
Description: Patient death attributable to AMR
Time Frame: Day 1 to Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 22
Participants | 1

11. Other Pre Specified Outcome: Non-lung Irreversible End-organ Failure
Description: Non-lung irreversible end-organ failure
Time Frame: Day 1 to Day 16
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 22
Participants | 1

12. Other Pre Specified Outcome: Incidence of Adverse Effects (AE)
Description: Incidence of adverse effects (AE)
Time Frame: Day 1 to Day 16
Population: Incidence of adverse effects (AE)
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 22
Participants | 22

13. Other Pre Specified Outcome: Incidence of Adverse Effects (AE) Requiring Dose-modification
Description: Incidence of adverse effects (AE) requiring dose-modification
Time Frame: Day 1 to Day 16
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 22
Participants | 5

14. Other Pre Specified Outcome: Incidence of Hypogammaglobulinemia
Description: Incidence of hypogammaglobulinemia
Time Frame: Day 1 to Day 16
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 22
Participants | 0

15. Other Pre Specified Outcome: Incidence of Culture-proven de Novo Infection
Description: Incidence of culture-proven de novo infection
Time Frame: Day 1 to Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 22
Participants | 6

16. Other Pre Specified Outcome: Diagnosis of Systemic Inflammatory Response Syndrome
Description: Diagnosis of systemic inflammatory response syndrome
Time Frame: Day 1 to Day 16
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 22
Participants | 0

17. Other Pre Specified Outcome: Patient Death
Description: Patient death
Time Frame: Day 1 to Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Treatment Arm
Number analyzed (Participants) | 22
Participants | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Carfilzomib Treatment Arm
All-Cause Mortality (participants affected / at risk) | 3/22
Serious Adverse Events (participants affected / at risk) | 4/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib Treatment Arm (N=22)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nervous system disorders - Other (Brain Herniation) (Nervous system disorders) | 1 (1) — brain herniation
diverticulitis with perforation (Gastrointestinal disorders) | 1 (1)
thombotic microangiopathy with acute renal failure (Renal and urinary disorders) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 1 (1) — Sepsis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib Treatment Arm (N=22)
Anemia (Blood and lymphatic system disorders) | 12 (18)
Acute kidney injury (Renal and urinary disorders) | 15 (24)
Bloating (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Confusion (Psychiatric disorders) | 1 (1)
Edema limbs (General disorders) | 6 (7)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Erythema
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Facial Tingling
Fatigue (General disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (10)
INR increased (Investigations) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
White blood cell decreased (Investigations) | 12 (22)
Lymphocyte count decreased (Investigations) | 12 (22)
Nausea (Gastrointestinal disorders) | 4 (8)
Neutrophil count decreased (Investigations) | 3 (4)
Platelet count decreased (Investigations) | 9 (13)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumonia
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT02474927/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT02474927/ICF_001.pdf